CLINICAL TRIAL: NCT01435642
Title: Diabcare Paediatric - A Survey-study on Diabetes Management, Complications and Psychosocial Aspects of Type 1 Childhood Diabetics
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Children With Type 1 Diabetes
Acronym: Diabcare
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3956; U1111-1122-1671 (Other: WHO)
Record Dates: First submitted 2011-08-31; First posted 2011-09-16 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will fill out a questionnaire when entering the non-interventional study

SUMMARY:
This study is conducted in Africa. The aim of this non-interventional study is to evaluate the current status of diabetes management, complications and psychosocial aspects for children with type 1 diabetes in Algeria.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the patient and his legal representative before any study-related activities (Study-related activities are any procedure related to recording of data according to the protocol)
* Type 1 diabetes
* Time since diabetes diagnosed at least 5 years
* Followed for diabetes at consultation for at least 12 months

Exclusion Criteria:

* Patient previously included in this study
* Secondary diabetes
* Pregnant patient
* Patient consulting for an emergency

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with type 1 diabetes mellitus being treated at diabetes clinics will be selected according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean HbA1c (glycosylated haemoglobin) | At the first visit (only one study visit) after 12 month of follow up

SECONDARY OUTCOMES:
Percentage of patients on insulin therapy | At the first visit (only one study visit) after 12 month of follow up
Mean duration of insulin therapy | At the first visit (only one study visit) after 12 month of follow up
Mean number of insulin injections/day | At the first visit (only one study visit) after 12 month of follow up
Mean insulin units per day | At the first visit (only one study visit) after 12 month of follow up
Percentage of patients on OAD or other treatments | At the first visit (only one study visit) after 12 month of follow up
Percentage of patients having complications (ophthalmological, peripheral, renal and others) | At the first visit (only one study visit) after 12 month of follow up
To quantify quality of life | At the first visit (only one study visit) after 12 month of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Blida, Algeria

REFERENCES:
- [Result] La prise en charge du diabéte de type 1 chez l'enfant en Algérie (DiabCare Pédiatrique); Bensenouci A, Achir M et al.; Médecine des Maladies Métaboliques 2015; Doi: 10.1016/S1957-2557(14)70902-2
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com